CLINICAL TRIAL: NCT03404245
Title: Empowering Active Self-management of Arthritis: Raising the Bar With OPERAS (an On-demand Program to EmpoweR Active Self-management)
Brief Title: an On-demand Program to EmpoweR Active Self-management (OPERAS)
Acronym: OPERAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Simon Fraser University (Other); Arthritis Research Centre of Canada (Other); Vancouver General Hospital (Other); The Arthritis Society, Canada (Other); Fraser Health (Other)
Responsible Party: Principal Investigator, Linda Li, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: H17-03424
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Joint Disease; Rheumatoid Arthritis
Keywords: Physical Activity; Exercise; Rheumatoid; Arthritis; Self-management; Symptoms
MeSH Terms: conditions — Joint Diseases; Arthritis, Rheumatoid; Motor Activity; Arthritis | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Active Comparator): Education, Fitbit/self-management web app, physiotherapist counselling. These 3 components will be delivered to the participants in Months 1 and 2. The session will include a short presentation about physical activity in everyday life, an individual goal-setting session with a registered physical therapist (PT), and an orientation to the Fitbit device and the web app. Participants will be provided access to a Fitbit and an app account. The PT will review physical activity goals with participants via bi-weekly phone calls and progressively modify their activities. In Month 3-6, participants will continue using Fitbit and the app and have access to a PT via email as needed, but no phone call. In Months 7-12, participants may keep their Fitbit and app account, but will not have access to a PT.
  Interventions: Behavioral: Education, Fitbit/self-management app, physiotherapist counselling.
- Delayed Intervention Group (Placebo Comparator): Same intervention with a 6 month delay: The full intervention will be initiated in Month 7 and 8 with a brief education session, use of a Fitbit paired with the self-management web app, and counseling by a physical therapist (PT). In Month 9-12, participants will continue the intervention without the PT phone calls, but will have email access to PT, if needed.
  Interventions: Behavioral: Same intervention with a 6 month delay

INTERVENTIONS:
Behavioral: Education, Fitbit/self-management app, physiotherapist counselling. — Participants will receive a brief education session, use a physical activity tracker Fitbit Flex paired with a self-management app, and remote counseling by a PT. Intervention will be received immediately.
  Arms: Immediate Intervention Group
Behavioral: Same intervention with a 6 month delay — The Delayed Intervention Group will receive the same intervention as the Immediate Intervention Group, but with a 6 month delay.
  Arms: Delayed Intervention Group

SUMMARY:
Self-management is a key component of successful chronic disease management and patients can benefit from learning about how daily activities and treatments relate to their symptoms and health status on an ongoing basis. The primary goal of this randomized controlled trial is to assess the efficacy of an e-health intervention, OPERAS, which includes two components: 1) the use of a newly developed web app to self-monitor symptoms/disease activity and treatment use, and help patients identify when a medical visit or treatment change is needed; 2) remote activity counselling provided by a physiotherapist, with the use of a wearable device (Fitbit) and the app to provide activity level feedback. The app component of OPERAS is hosted by the secure network of Arthritis Research Canada.

DETAILED DESCRIPTION:
Self-management is a fundamental component in arthritis care, however, it is often neglected as most models of arthritis care focus on early access to medical consultation and surgical interventions. Patient self-management refers to the active participation of patients in a variety of activities that contribute to lessening the physical and emotional impact of illnesses. There are several factors attributing to a lack of self-management practice, such as frustration from managing health on a trial-and-error basis, a lack of knowledge to effectively monitor symptoms and disease, and being unsure about how to manage physical activities without aggravating symptoms. The variety of risk factors highlight the need for a multifaceted approach that provides support in terms of knowledge, skill development and timely advice from health professionals, as well as motivational support for patients to be engaged in their care and to stay physically active.

Our primary objective is to assess the efficacy of an e-health intervention, OPERAS, which integrates the Arthritis Health Journal and a Physical Activity Counselling program, to improve self-management ability. Our secondary objectives are to explore the effect of the intervention on disease status and physical activity levels and to assess barriers to implementation and sustainability of the e-health intervention in (rheumatoid arthritis) RA management.

The investigators will use a mixed-methods approach, involving a randomized controlled trial (RCT) and in-depth interviews. The proof-of-concept study will employ a stepped wedge RCT design, whereby the intervention will be sequentially rolled out to participants over a number of time periods. The order in which individuals receive the intervention will be determined at random. The strength of this design is that it can properly address the efficacy question, while avoiding the dilemma of withholding the intervention to some participants, as in a parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* a physician confirmed diagnosis of RA
* no joint surgery in the past 6 months
* no history of acute injury to any joints in the past 6 months
* an email address and daily access to a computer or mobile device.

Exclusion Criteria:

* people who should not be physically active without medical supervision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure | Baseline
  Patient Activation Measure is a 13-item self-reported measure of individuals' confidence in managing chronic diseases. Each item has a 4-point response (1 "strongly disagree"; 4 "strongly agree"), with the aggregate raw score converted to 0-100. Hibbard et al presented a 4-stage activation model derived from the standardized scores: 1) Believing an active role is important (PAM score <47); 2) Having confidence and knowledge to take action (47.1 - 55.1); 3) Taking action (55.2 - 67); 4) Maintaining healthy behaviours despite setbacks (> 67.1).
Patient Activation Measure | 6 months
  Patient Activation Measure is a 13-item self-reported measure of individuals' confidence in managing chronic diseases. Each item has a 4-point response (1 "strongly disagree"; 4 "strongly agree"), with the aggregate raw score converted to 0-100. Hibbard et al presented a 4-stage activation model derived from the standardized scores: 1) Believing an active role is important (PAM score <47); 2) Having confidence and knowledge to take action (47.1 - 55.1); 3) Taking action (55.2 - 67); 4) Maintaining healthy behaviours despite setbacks (> 67.1).
Patient Activation Measure | 12 months
  Patient Activation Measure is a 13-item self-reported measure of individuals' confidence in managing chronic diseases. Each item has a 4-point response (1 "strongly disagree"; 4 "strongly agree"), with the aggregate raw score converted to 0-100. Hibbard et al presented a 4-stage activation model derived from the standardized scores: 1) Believing an active role is important (PAM score <47); 2) Having confidence and knowledge to take action (47.1 - 55.1); 3) Taking action (55.2 - 67); 4) Maintaining healthy behaviours despite setbacks (> 67.1).

SECONDARY OUTCOMES:
Rheumatoid Arthritis Disease Activity Index | Baseline
  Rheumatoid Arthritis Disease Activity Index consists of: 1) global disease activity; 2) joint tenderness/swelling; 3) pain; 4) morning stiffness; 5) number/severity of painful joints. Score ranges from 0 - 10; lower = better.
Rheumatoid Arthritis Disease Activity Index | 6 months
  Rheumatoid Arthritis Disease Activity Index consists of: 1) global disease activity; 2) joint tenderness/swelling; 3) pain; 4) morning stiffness; 5) number/severity of painful joints. Score ranges from 0 - 10; lower = better.
Rheumatoid Arthritis Disease Activity Index | 12 months
  Rheumatoid Arthritis Disease Activity Index consists of: 1) global disease activity; 2) joint tenderness/swelling; 3) pain; 4) morning stiffness; 5) number/severity of painful joints. Score ranges from 0 - 10; lower = better.
Daily Moderate/Vigorous Physical Activity time | Baseline
  Time spent in Moderate/Vigorous Physical Activity (MVPA) is measured with a SenseWear Mini sensor over a 7-day period. We will calculate the mean time spent in bouted MVPA per day. A bout is defined as >= 10 consecutive minutes or more at the level of >= 3 METs (i.e., the lower bound of MVPA), with allowance for interruption of up to one minute below the threshold.
Daily Moderate/Vigorous Physical Activity time | 6 months
  Time spent in Moderate/Vigorous Physical Activity (MVPA) is measured with a SenseWear Mini sensor over a 7-day period. We will calculate the mean time spent in bouted MVPA per day. A bout is defined as >= 10 consecutive minutes or more at the level of >= 3 METs (i.e., the lower bound of MVPA), with allowance for interruption of up to one minute below the threshold.
Daily Moderate/Vigorous Physical Activity time | 12 months
  Time spent in Moderate/Vigorous Physical Activity (MVPA) is measured with a SenseWear Mini sensor over a 7-day period. We will calculate the mean time spent in bouted MVPA per day. A bout is defined as >= 10 consecutive minutes at the level of >= 3 METs (i.e., the lower bound of MVPA), with allowance for interruption of up to one minute below the threshold.
Daily sedentary time | Baseline
  Time spent in sedentary activity is measured with a SenseWear Mini sensor over a 7-day period. We will calculate the mean daily time spent in sedentary activity, with an energy expenditure of <=1.5 METs, occurring in bouts of >= 20 minutes during waking hours
Daily sedentary time | 6 months
  Time spent in sedentary activity is measured with a SenseWear Mini sensor over a 7-day period. We will calculate the mean daily time spent in sedentary activity, with an energy expenditure of <=1.5 METs, occurring in bouts of >= 20 minutes during waking hours
Daily sedentary time | 12 months
  Time spent in sedentary activity is measured with a SenseWear Mini sensor over a 7-day period. We will calculate the mean daily time spent in sedentary activity, with an energy expenditure of <=1.5 METs, occurring in bouts of >= 20 minutes during waking hours

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PhD, Principal Investigator — Professor
Locations (1):
- Arthritis Research Canada, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feehan L, Xie H, Lu N, Li LC. Twenty-four hour physical activity, sedentary behaviour and sleep profiles in adults living with rheumatoid arthritis: a cross-sectional latent class analysis. J Act Sedentary Sleep Behav. 2024 Apr 17;3(1):10. doi: 10.1186/s44167-024-00049-5. PMID 40217417
- [Derived] Tam J, Lacaille D, Liu-Ambrose T, Shaw C, Xie H, Backman CL, Esdaile JM, Miller K, Petrella R, Li LC. Effectiveness of an online self-management tool, OPERAS (an On-demand Program to EmpoweR Active Self-management), for people with rheumatoid arthritis: a research protocol. Trials. 2019 Dec 11;20(1):712. doi: 10.1186/s13063-019-3851-0. PMID 31829286